CLINICAL TRIAL: NCT03268551
Title: Does Medical Cannabis Reduce Opioid Analgesics in HIV+ and HIV- Adults With Pain?
Brief Title: MEMO-Medical Marijuana and Opioids Study
Status: Completed | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Fordham University (Other); Columbia University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2017-7857; 1R01DA044171-01A1 (NIH)
Record Dates: First submitted 2017-08-23; First posted 2017-08-31 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Opioid Use; Marijuana; Chronic Pain; HIV/AIDS
MeSH Terms: conditions — Marijuana Abuse; Chronic Pain; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will examine how medical cannabis use affects opioid analgesic use over time, with particular attention to THC/CBD content, HIV outcomes, and severe adverse events.

DETAILED DESCRIPTION:
The overarching goal of the study is to understand how medical cannabis use affects opioid analgesic use over time, with particular attention to THC/CBD content, HIV outcomes, and adverse events. The study will include a cohort of 250 HIV+ and HIV- adults with (a) severe or chronic pain, (b) opioid analgesic use, and (c) new certification for medical cannabis. Over 18 months, participants will have 7 in-person visits every 3 months and 39 web-based questionnaires every 2 weeks. Data sources will include questionnaires; medical, pharmacy, and Prescription Monitoring Program records; and urine and blood samples. Over each 2-week time period (unit of analysis), the primary exposure measure will be number of days of medical cannabis use, and the primary outcome measure will be cumulative opioid analgesic dose. Qualitative interviews will also be conducted with a subgroup of 30 participants to explore perceptions of how medical cannabis use affects opioid analgesic use. Qualitative findings will help understand the reasons underlying the findings of the cohort study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* English or Spanish fluency
* New certification for medical cannabis within 90 days
* No medical cannabis use in the 6 months prior to certification
* Medical cannabis qualifying complication of "chronic or severe pain"
* Use of prescribed or illicit opioid analgesics within 30 days

Exclusion Criteria:

* Inability to provide informed consent
* Inability to complete study visits over 18 months
* Qualifying conditions for medical cannabis in NY that are likely to cause unique pain syndromes (cancer, epilepsy, multiple sclerosis, spinal cord injury, amyotrophic lateral sclerosis, Parkinson's disease, inflammatory bowel disease, Hungtington's disease)
* Terminal illness
* Current or prior psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with chronic pain, who are taking opioids, and who are newly certified for medical marijuana in NY.
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Opioid analgesic use | Opioid analgesic use will be a cumulative dose of all opioid analgesics over each of the 39 2-week periods.
  The primary outcome will combine measures of prescribed and illicit opioid analgesic use.

SECONDARY OUTCOMES:
Alternative measures of opioid analgesic use | Alternative measures of opioid analgesic use will be measured over each of the 39 2-week periods.
  Alternative measures of opioid analgesic use will include: number of days of all opioid analgesic use, mean daily dose of all opioid analgesics, cumulative dose of prescribed (only) opioid analgesics, number of days of prescribed (only) opioid analgesic use, and mean daily dose of prescribed (only) opioid analgesic use.
HIV viral load | HIV outcomes will be measured seven times every 3 months from baseline through 18 months.
  HIV viral load will be measured in copies/ml from blood samples collected during the study.
CD4 count | CD4 count will be measured seven times every 6 months from baseline through 18 months..
  CD4 count will be measured in cells/mm3 from blood samples collected during the study.
HIV antiretroviral adherence | HIV antiretroviral adherence will be measured seven times every 3 months from baseline through 18 months..
  HIV antiretroviral adherence will be a composite measure from self-reported questionnaires and pharmacy records.
HIV risk behaviors | HIV risk behaviors will be measured seven times every 3 months from baseline through 18 months..
  HIV risk behaviors will be a composite measure from self-reported questionnaires.
Cannabis use disorder | Cannabis use disorder will be measured three times every 6 months.
  Cannabis use disorder will be measured using standardized instruments.
Illicit drug use | Illicit drug use will be measured seven times every 3 months from baseline through 18 months..
  Illicit drug use will be measured using standardized surveys and urine toxicology testing.
Diversion of medical cannabis | Diversion will be measured seven times every 3 months from baseline through 18 months..
  Diversion will be measured using standardized surveys.
Non-fatal overdose | Non-fatal overdose will be measured seven times every 3 months from baseline through 18 months..
  Non-fatal overdose will be measured using standardized surveys.
Death | Death will be measured 18 months after enrollment.
  Death will be ascertained from the National Death Index
Accidents/Injuries | Accident/Injuries will be measured seven times every 3 months from baseline through 18 months..
  Accidents/Injuries will be measured using standardized survey instruments

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Montefiore Health System, The Bronx, New York
  - Vireo Health, White Plains, New York

REFERENCES:
- [Derived] Zhang C, Slawek DE, Ross J, Zolotov Y, Castillo F, Levin FR, Sohler NL, Minami H, Cunningham CO, Starrels JL, Arnsten JH. Factors Associated with Medical Cannabis Use After Certification: A Three-Month Longitudinal Study. Cannabis Cannabinoid Res. 2024 Jun;9(3):e859-e869. doi: 10.1089/can.2022.0248. Epub 2023 Mar 24. PMID 36961410
- [Derived] Cunningham CO, Starrels JL, Zhang C, Bachhuber MA, Sohler NL, Levin FR, Minami H, Slawek DE, Arnsten JH. Medical Marijuana and Opioids (MEMO) Study: protocol of a longitudinal cohort study to examine if medical cannabis reduces opioid use among adults with chronic pain. BMJ Open. 2020 Dec 29;10(12):e043400. doi: 10.1136/bmjopen-2020-043400. PMID 33376181
- See also: Medical Marijuana and Opioids (MEMO) Study: protocol of a longitudinal cohort study to examine if medical cannabis reduces opioid use among adults with chronic pain — https://bmjopen.bmj.com/content/10/12/e043400
- See also: Pain catastrophizing and mental health phenotypes in adults with refractory chronic pain: A latent class analysis — https://doi.org/10.1016/j.jpsychires.2021.12.001